CLINICAL TRIAL: NCT03175601
Title: Sleep Disturbances and Biomarkers of Sarcopenic OBesity: Insight Into Mechanisms of Prefrailty
Brief Title: Sleep Disturbances and Biomarkers of Sarcopenic OBesity
Acronym: SleSOB
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Istituto di Fisiologia Clinica CNR (Other)
Collaborators: Niguarda Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 422-102016
Record Dates: First submitted 2017-06-01; First posted 2017-06-05 (Actual); Last update posted 2017-06-06 (Actual); Status verified 2017-06

CONDITIONS: Sarcopenic Obesity
Keywords: Sleep disturbances; Biomarkers; Prefrailty; Insulin resistance; Olfactory impairment; Multiplex array; Gait speed
MeSH Terms: conditions — Parasomnias; Insulin Resistance; Olfaction Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Serum, plasma and urine samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The general objective of this study is to identify biomarkers of sleep quality, sarcopenia, insulin resistance, oxidative stress and inflammation associated with prefrailty in middle-aged and elderly obese subjects through the integrated study of sleep patterns, functional cardiovascular testing, olfactory function and circulating molecules.

Results from the SleSOB study will contribute to identify molecular and functional determinants of prefrailty, to allow early targeted interventions and will have important implications for empowerment of elderly citizens to self-management of preventive measures and healthy lifestyle.

DETAILED DESCRIPTION:
Frailty, an age-related state of low physiological reserve and high vulnerability to stressors, impacts on health, functional independence, quality of life and survival; its early detection at the prefrailty stage offers the opportunity for preventive intervention. Sarcopenia, a hallmark of frailty, may occur in association with obesity and worsen functional deterioration. Obesity is strongly associated with insulin resistance and is a risk factor for both cardiometabolic diseases and cognitive impairment. Adipose tissue exerts autocrine and paracrine functions leading to chronic low-grade inflammation and increased oxidative stress that, in turn, decrease muscle density and precipitate muscle strength loss. Sleep disturbances and sarcopenia might be causally related through dysregulation of glucose metabolism and disruption of the secretory pattern of hormones involved in muscle metabolism.

Main objective:

To establish among young-elderly obese subjects the prevalence of prefrailty as defined by presence of ≥1 of reduced muscle mass, fatigue, weakness, slowness, and low physical activity (Fried's criteria)

Secondary objectives:

* To assess prevalence and severity of sarcopenia as defined by reduced muscle mass coupled with decreased muscle strength and /or reduced functional capacity
* To establish the cardiometabolic risk profile and its correlation with vitamin D
* To determine type and extent of sleep abnormalities by validated questionnaires and their association with prefrailty
* To assess the extent of sympathetic imbalance, arrhythmia burden and olfactory impairment
* To determine patterns of biomarkers of oxidative stress, inflammatory cytokines, adipokines, myokines, tissue damage and remodeling and correlation with prefrailty and insulin resistance.

Study design:

Eligible subjects will attend the clinic in the morning in the fasting state to undergo

* blood samples collection for routine and specific biochemistry;
* anthropometric measurements: height, weight, body mass index, waist and hip circumference;
* assement of sarcopenia: muscle strength, gait speed, muscle mass by biomimpedentiometric assessment (BIA) and air displacement pletismography (BODPOD);
* glucose metabolism biomarker as tissue accumulation of advanced glycation endproducts (AGE);
* sympathetic activation;
* interview for medical history and comorbidity registration;
* screening for cognitive impairment;
* sleep pattern analysis through questionnaires;
* olfactory assessment.

A wearable system (Win@home, CE0434) for 24 h recording of rhythm, circadian heart rate, respiratory rate and oxygen saturation, posture and physical activity will be applied to each subject for the subsequent 24 hours

ELIGIBILITY:
Inclusion Criteria:

* Obesity : body mass index ≥ 30 and <40 kg/m2
* Written informed consent

Exclusion Criteria:

* Diabetes requiring insulin treatment
* Stage IV chronic kidney dysfunction (estimated glomerular filtration rate <15 ml/min)
* Liver dysfunction (AST- ALT x 2 times upper normalcy range)
* Active neoplasms
* Claustrophobia
* Psychiatric morbidity or any other condition that impairs the ability to give informed consent

Ages: 55 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Middle-aged and young-old obese subjects will be enrolled at a specialised nutrition clinic. Subjects will be on a maintenance weight management program including lifestyle advice and diet based on the principles of the Modern Mediterranean Diet Pyramid (variety in food choices, seasonality and spices to flavor dishes). The diet is modified to avoid high caloric food and distributed in 3 main meals and 2 healthy snacks during the day to provide a caloric intake of 28-30 kcal/die/kg body weight and macronutrient breakdown as recommended by INRAN (http://www.inran.it/) (Protein 15%, Fat < 30%, carbohydrates 55/60% of which soluble 10-12 % and fiber 30 g die).
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-06 (Estimated); Primary Completion 2018-05 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Prevalence of prefrailty | Day one
  Proportion of subjects presenting with one or more of reduced muscle mass, fatigue, weakness, slowness, and low physical activity

SECONDARY OUTCOMES:
Prevalence of sarcopenia | Day one
  Proportion of subjects presenting with reduced muscle mass (by gender-specific cut offs ) coupled with decreased muscle strength (men ≤ 32 kg, women ≤ 21 kg and/or reduced gait speed (<0.8 mt/sec on a 4 mt course)
Cardiometabolic risk profile: insulin resistance | Day one
  Homeostatic Model Assessmenti (HOMA)-insulin resistance index
Cardiometabolic risk profile: fatty liver | Day one
  Fatty liver index (FLI)
Cardiometabolic risk profile: 10-year cardiovascular risk | Day one
  HeartSCORE
Sleep abnormalities: idiopathic REM Behaviour Disorder (iRBD) | Day one
  Answer to screening question for iRBD
Sleep abnormalities: insomnia severity | Day one
  Insomnia Severity Index (ISI) score
Sleep abnormalities: daytime sleepiness | Day one
  Epworth Sleepiness Scale (ESS) score
Cardiac rhythm abnormalities | Day one
  Atrial fibrillation burden during 24 hour home monitoring
Cardiac dysautonomia: deep breathing test | Day one
  Expiratory/inspiratory ratio
Cardiac dysautonomia: lying to standing test | Day one
  Lying-to standing ratio
Orthostatic hypotension | Day one
  Drop ≥20 mmHg in systolic and/or ≥10 mmHg in diastolic blood pressure after 1 and 5 minutes of active standing
Olfactory function: Total Olfactory Score (TOS) | Day one
  Sum of Olfactory Threshold, Identification, Discrimination scores
Screening for cognitive impairment | Day one
  Mini Mental State Examination (MMSE) score
Tissue accumulation of Advanced Glycation End-products (AGE) | Day one
  AGE Reader Score
Biomarkers of oxidative stress | Day one
  Malondyaldehyde, aminothiols
Inflammatory biomarkers | Day one
  Cytokinesinterleukin-6, interleukin-1beta, tumour ecrosis Factor-alpha, neopterin
Adipokines | Day one
  Adiponectin, leptin
Myokines | Day one
  Myostatin, irisin

CONTACTS AND LOCATIONS:
Overall Officials: Maria Giovanna Trivella, MD, Principal Investigator — Istituto di Fisiologia Clinica CNR; Jonica Campolo, MSc, Study Director — Istituto di Fisiologia Clinica CNR
Locations (1):
- Istituto di Fisiologia Clinica del CNR UOS Milano, Milan, Italy

IPD SHARING:
Plan to Share IPD: No